CLINICAL TRIAL: NCT04355013
Title: Temperature Monitoring in Cardiac Surgery: Clinical Study of Agreement Between Different Measurement Methods
Brief Title: Temperature Monitoring in Cardiac Surgery: Agreement Between Different Clinical Methods
Status: Completed | Type: Observational
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Responsible Party: Principal Investigator, Jose Alfonso Sastre, Principal investigator, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Other Study IDs: CAUSA27/04/2016
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Temperature Change, Body
Keywords: Core temperature; Cardiac surgery
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Core emperature monitoring — Monitoring core temperatures with probes placed in the arterial outlet and venous inlet of extracorporeal pump, pulmonary artery, bladder, nasopharinx and forehead using a doublé-sensor probe

SUMMARY:
Observational study to compare core temperatures obtained by 6 methods in patients undergoing cardiac surgery under cardiopulmonary bypass.

DETAILED DESCRIPTION:
This study compares the core temperatures obtained by means of different probes placed in nasopharinx, pulmonary artery, arterial outlet, venous inlet, bladder and forehead in patients undergoing cardiac surgery under cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Only patients requiring a pulmonary artery catheter were included.

Exclusion Criteria:

* Sepsis or previous fever.
* Previous bladder catheter without termistor
* Deep hypothermic circulatory arrest.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery under cardiovascular bypass
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-09-28; Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IBSAL, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sastre JA, Lopez T, Moreno-Rodriguez MA, Reta-Ajo L, Rubia-Martin MC, Diez-Castro R. Reliability of different body temperature measurement sites during normothermic cardiac surgery. Perfusion. 2023 Apr;38(3):580-590. doi: 10.1177/02676591211069918. Epub 2022 Feb 8. PMID 35133212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients undergoing cardiac surgery using cardiopulmonary bypass and requiring hemodynamic monitoring by means of a pulmonary artery catheter.
Pre-assignment Details: Exclusion criteria were sepsis or previous fever, presence of a previous standard urinary bladder catheter (without thermistor) inserted prior to surgery, moderate hypothermic cardiopulmonary bypass, or deep hypothermic circulatory arrest.
Groups:
- Patients Undergoing CPB Cardiac Surgery.: Adult patients undergoing cardiac surgery using cardiopulmonary bypass and requiring hemodynamic monitoring by means of a pulmonary artery catheter.
Period: Overall Study
Arm/Group | Patients Undergoing CPB Cardiac Surgery.
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing CPB Cardiac Surgery.
Number analyzed (Participants) | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Median (Inter-Quartile Range); unit: kilograms] | 70 [64 to 82]
Height [Median (Inter-Quartile Range); unit: centimeters] | 165 [160 to 170]

OUTCOME MEASURES:

1. Primary Outcome: Agreement Between Different Core Temperature Methods
Description: Agreement between core temperatures obtained in arterial CPB output versus venous inlet of CPB, bladder, pulmonary artery, nasopharynx and forehead (Tcore). The measurements were compared between the different methods using the Bland-Altman method of repeated measures and expressed as mean difference (reference method-alternative method) plus CI95%.
Time Frame: 24 temperature measures per patient recorded at 5-min intervals for each method and averaged using the Bland-Altman method for repeated measures
Measure: Median (95% Confidence Interval); unit: celsius degrees (mean difference)
Groups:
- Arterial Outlet: Temperature in CPB arterial outlet
- Nasopharyngeal: Temperature in nasopharynx
- Bladder: Temperature in bladder
- Tcore: Skin temperature measure with Tcore
- Venous Inflow: CPB venous inflow temperature
Arm/Group | Arterial Outlet | Nasopharyngeal | Bladder | Tcore | Venous Inflow
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
celsius degrees (mean difference) | 35.0 [34.9 to 35.0] | 35.2 [35.1 to 35.3] | 35.6 [35.5 to 35.6] | 34.8 [34.7 to 35.0] | 34.8 [34.7 to 34.9]
Statistical Analysis 1: Comparison: Arterial Outlet vs Nasopharyngeal; Arterial outlet-nasopharyngeal temperatures; Test type: Other — Agreement between different methods of temperature measurement (Bland-Altman plot with multiple measurements per individual); Bland-Altman for repeated measures = -0.16, 95% CI 2-sided [-1.10 to 0.77], Standard Deviation 0.47
Statistical Analysis 2: Comparison: Arterial Outlet vs Venous Inflow; Arterial-venous inflow temperatures; Test type: Other — [test comment as in outcome 1, analysis 1]; Bland-Altman; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.63 to 0.95], Standard Deviation 0.4
Statistical Analysis 3: Comparison: Arterial Outlet vs Bladder; Arterial outlet-bladder; Test type: Other — [test comment as in outcome 1, analysis 1]; Bland-Altman; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.98 to 0.74], Standard Deviation 0.69
Statistical Analysis 4: Comparison: Arterial Outlet vs Tcore; Arterial outlet- Tcore; Test type: Other — [test comment as in outcome 1, analysis 1]; Bland-Altman; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-1.38 to 1.54], Standard Deviation 0.74
Statistical Analysis 5: Comparison: Nasopharyngeal vs Venous Inflow; Nasopharyngeal-venous inflow temperatures; Test type: Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.73 to 1.38], Standard Deviation 0.53
Statistical Analysis 6: Comparison: Nasopharyngeal vs Bladder; Nasopharyngeal-bladder temperatures; Test type: Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.50 to 0.59], Standard Deviation 0.52
Statistical Analysis 7: Comparison: Nasopharyngeal vs Tcore; Nasopharyngeal-Tcore temperatures; Test type: Other — Bland-Altman for repeated measures; Bland-Altman for repeated measures = 0.24, 95% CI 2-sided [-0.90 to 1.39], Standard Deviation 0.58

ADVERSE EVENTS:
Time Frame: No adverse effects were measured
Description: It is an observational study comparing different methods of temperature monitoring in cardiac surgery
Groups:
- No Adverse Effects Were Measured: No adverse effects were measured
Arm/Group | No Adverse Effects Were Measured
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT04355013/Prot_SAP_000.pdf